CLINICAL TRIAL: NCT04974281
Title: Efficacy and Safety of PD-1 Antibody and Lenvatinib Plus TACE on Downstaging Hepatocellular Carcinoma With BCLC B/C
Brief Title: PD-1 Antibody and Lenvatinib Plus TACE on Downstaging BCLC B/C HCC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Director, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUASHAN007
Record Dates: First submitted 2021-06-20; First posted 2021-07-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Lenvatinib; PD-1; TACE; Downstaging
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1+TACE+Len (Other): PD-1 Antibody and Lenvatinib Plus TACE
  Interventions: Combination Product: PD-1 and Lenvatinib Plus TACE

INTERVENTIONS:
Combination Product: PD-1 and Lenvatinib Plus TACE — PD-1 Antibody and Lenvatinib Plus Transarterial chemoembolization(TACE )： Patients were recommended to receive TACE once every 6 weeks. Patients were recommended to begin oral administration of Lenvatinib 3 days after the first TACE treatment, and meanwhile to start intravenous drip of PD-1 antibody 3 days after the first TACE treatment, once every 3 weeks.

SUMMARY:
The purpose of this study is to assess the difference of safety and efficacy about PD-1 Antibody and Lenvatinib Plus transcatheter arterial chemoembolization (TACE) on downstaging hepatocellular carcinoma with BCLC B/C.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old;
2. Clinically diagnosed as hepatocellular carcinoma, stage B/C of BCLC;
3. No history of severe arrhythmia or heart failure;
4. No history of severe ventilation dysfunction or severe pulmonary infection;
5. No acute or chronic renal failure, the creatinine clearance rate was >40 mL/min;
6. Liver function Child A;
7. Blood routine: absolute neutrophils count ≥1.5×10^9/L, Hb≥8.5g/L, PLT≥75×10^9/L;
8. Coagulation function: INR≤2.3;
9. ECOG score <2;
10. No local or systemic treatment, such as TACE, RFA, targeted drugs, traditional Chinese medicine, etc., before enrollment;
11. Expected survival ≥12 weeks;
12. At least one lesion can be measured and evaluated by CT/MRI according to RECIST 1.1 criteria;
13. Understand and sign the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with other malignant tumors;
3. patients with complicated mental illness;
4. patients who have participated in other clinical trials in the last three months;
5. known or suspected allergy to any drug related to the study;
6. Patients with positive immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
7. Patients treated with other targeted drugs, PD-L1 antibody and other immunotherapy or FOLFOX systemic chemotherapy after inclusion;
8. Patients with ≥1 + proteinuria indicated by urine routine will receive 24-hour urine protein detection, and patients with ≥1g 24-hour urine protein will not be included in the group.
9. Active autoimmune diseases that require systemic treatment (use of disease-alleviating agents, such as corticosteroids or immunosuppressants)
10. Patients with uncontrolled hepatitis B/C infection
11. Other conditions that the researcher considers not suitable for inclusion in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Resection rate | 6 months after downstaging treatment
  Resction rate refers to the proportion of patients who can receive radical surgery after downstaging treatment.

SECONDARY OUTCOMES:
Adverse events (safety) | 6 months
  Postoperative adverse events (safety ) will be evaluated according to the NCI CTCAE Version 4.03.The number and severity of treatment-related side effects, including AE and SAE, will be recorded during treatment.
Overall survival (OS) | 2 years
  The duration from the date of recruitment to the date of death from any cause.
Objective response rate (ORR) | 6 months
  ORR is defined as the percentage of participants who have a confirmed complete response or partial response according to RECIST 1.1 or mRECIST.
Progression free survival (PFS) | 6 months
  PFS is defined as the time from enrollment of the trial to the first documented disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Lunxiu Qin, M.D, Study Director — Department of Surgery, Huashan Hospital, Fudan University
Locations (1):
- Huashan hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Lencioni R, de Baere T, Soulen MC, Rilling WS, Geschwind JF. Lipiodol transarterial chemoembolization for hepatocellular carcinoma: A systematic review of efficacy and safety data. Hepatology. 2016 Jul;64(1):106-16. doi: 10.1002/hep.28453. Epub 2016 Mar 7. PMID 26765068
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Kato Y, Tabata K, Kimura T, Yachie-Kinoshita A, Ozawa Y, Yamada K, Ito J, Tachino S, Hori Y, Matsuki M, Matsuoka Y, Ghosh S, Kitano H, Nomoto K, Matsui J, Funahashi Y. Lenvatinib plus anti-PD-1 antibody combination treatment activates CD8+ T cells through reduction of tumor-associated macrophage and activation of the interferon pathway. PLoS One. 2019 Feb 27;14(2):e0212513. doi: 10.1371/journal.pone.0212513. eCollection 2019. PMID 30811474
- [Background] Kudo M, Ueshima K, Ikeda M, Torimura T, Tanabe N, Aikata H, Izumi N, Yamasaki T, Nojiri S, Hino K, Tsumura H, Kuzuya T, Isoda N, Yasui K, Aino H, Ido A, Kawabe N, Nakao K, Wada Y, Yokosuka O, Yoshimura K, Okusaka T, Furuse J, Kokudo N, Okita K, Johnson PJ, Arai Y; TACTICS study group. Randomised, multicentre prospective trial of transarterial chemoembolisation (TACE) plus sorafenib as compared with TACE alone in patients with hepatocellular carcinoma: TACTICS trial. Gut. 2020 Aug;69(8):1492-1501. doi: 10.1136/gutjnl-2019-318934. Epub 2019 Dec 4. PMID 31801872